CLINICAL TRIAL: NCT04553445
Title: Temporal, Environmental, and Genetic Factors Regulating Exercise and Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1607166
Record Dates: First submitted 2020-09-02; First posted 2020-09-17 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Migraine Disorders
Keywords: Chronotype; Green exercise
MeSH Terms: conditions — Migraine Disorders | interventions — Chronotype

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronotype (Experimental): Determination whether monthly migraine load is affected by exercise in sync with chronotype
  Interventions: Behavioral: Chronotype
- Green exercise (Experimental): Determination whether monthly migraine load is affected by exercise in a natural environment
  Interventions: Behavioral: Green exercise

INTERVENTIONS:
Behavioral: Chronotype — Participants screened using the Morningness/Eveningness Questionnaire. Chronotype categorized as either Definite Morning/Morning, or Evening/Definite Evening. Participant will exercise (60-70% estimated heart rate max, 2 x per week, 30-min/session) either in sync or not in sync with chronotype for one month in a randomized cross-over design. There will be a one-month wash out period, and then participant will complete training in the alternate chronotype for one month.
  Arms: Chronotype
Behavioral: Green exercise — Participants will be randomly assigned to four weeks of moderate intensity aerobic exercise (60-70% estimated heart rate max, 2 x per week, 30-min/session) in either natural or indoor environments in a randomized cross-over design. There will be a one-month wash out period, and then participant will complete training in alternate environment for one month.
  Arms: Green exercise

SUMMARY:
Chronic pain, of which migraine is among the most common, affects 100 million US adults and costs between $560 to $635 billion dollars annually. There is a need for effective, low-cost non-pharmacological strategies to reduce migraine load in migraineurs (based on International Headache Society classification International Classification of Headache Disorders [ICHD]-3; experience headache [migraine-like or tension-type-like] on 15+ days/month for 3+ months, and have migraine headaches [either with aura or without aura] on 8+ days/month). This represents an area of interest, as common migraine medications induce central nervous system side-effects including aphasia, ataxia, somnolescence, and vertigo; and 79% of suffers have an interest in trying novel treatment strategies with lower adverse effects than medications.

Exercise has been shown to be a non-pharmacological intervention to reduce migraine burden. However, how environmental (i.e. - time-of-day, exposure to nature) and genetic factors (i.e. - polymorphisms in circadian and migraine associated genes) impact the laudatory effects of exercise remains unknown. There are independently established heritable components to migraine frequency (65%), circadian rhythm (70%), and aerobic power during exercise (66%). Thus, the central hypothesis is that an optimal environment can improve the exercise-induced reduction in migraine load, which is influenced by genetic heritability of migraine related gene polymorphisms.

DETAILED DESCRIPTION:
Willing participants who are self-reported chronic migraineurs will complete an informed consent followed by a health risk questionnaire to determine study eligibility.

Phase I: Chronic migraineurs will be screened using the Morningness/Eveningness Questionnaire (MEQ) to recruit a cohort of discrepant chronotypes (Definite Morning, Morning; and Evening, Definite Evening). Resulting participants will be complete a baseline migraine load evaluation and assigned to four weeks of moderate intensity exercise (60-70% estimated heart rate max, 2 x per week, 30-min/session) consolidated to either the morning (before 09:00) or afternoon (after 17:00) in a randomized cross-over design. Intensity will be tracked through a heart rate monitor that will be provided to participants, and an application that they can download to their phone. Participants will be able to keep the heart rate monitor upon completion of the study. An example of potential exercises will be provided to participants and research team members will check in every 1-2 weeks to see how exercise is progressing. Migraine burden will be assessed pre- and post-training after each condition using the Migraine Disability Assessment (MIDAS) and the short version of the Headache Impact Test (HIT-6). Half of the participants will exercise for one month during a time of day that is in sync with their chronotype (i.e. Morning type person will exercise in the morning), and the other half of the participants will exercise at a time of day that is not in sync (i.e. Morning type person will exercise in the evening). There will be a one-month wash out period, and then participants will complete training at the other time of day. A buccal swab will be obtained (according to protocols outlined on our approved Institutional Biosafety Committee protocol) for phenotyping of genes specific to chronotype and migraine.

Phase II will also recruit chronic ICHD-3 migraineurs. Participants will complete a baseline migraine load evaluation as described above. If an effect of chronotype is found in Phase I, participants will complete exercise training in sync with their chronotype. Participants will be randomly assigned to four weeks of moderate intensity aerobic exercise (60-70% estimated heart rate max, 2 x per week, 30-min/session) in either natural or indoor environments in a randomized cross-over design. Intensity will be tracked through a heart rate monitor that will be provided to participants, and an application that they can download to their phone. Participants will be able to keep the heart rate monitor upon completion of the study. An example of potential exercises will be provided to participants and research team members will check in every 1-2 weeks to see how exercise is progressing. A recent investigation provided evidence that activity performed in a desert environment provided the same benefits as in a green landscape with respect to both cardiovascular measures as well as perception of comfort, calm, and perceived stress. Half of the participants will exercise for one month in a natural environment that they select (outdoors in a park, or trail) and the other half will complete exercise indoors (participants will not require access to fitness facilities, although these could be used if they are already a member). There will be a one month wash out period, and then participants will complete exercise training in the other setting. Change in the monthly migraine load will be determined between environments. A buccal swab will be obtained for phenotyping of genes specific to chronotype and migraine.

Buccal swab samples will be used to isolate DNA. Isolated DNA will be genotyped at the University of Nevada, Las Vegas (UNLV) Genomics Core Facility using polymerase chain reaction and then disposed of. Genotypes will be linked to participant migraine load responses, and then reported in aggregate.

The investigators plan to maintain regular contact with participants. After each exercise bout, participants will download and email the associated csv file which will be received, deidentified, and labelled with the participant identification number for digital storage at UNLV. In response, participants will be asked about the exercise sessions (with open ended questions such as "How do you feel the exercise sessions are going?"). The file will be reviewed upon receipt by a member of the research team to determine exercise intensity (60-70% estimated heart rate range), allow the investigators to provide feedback, and also enable the determination of how well participants are adhering to the intervention. The investigators will use the Polar Flow application (available for free), which can be deleted by the participant at the end of the study if they so choose.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be classified as a chronic migraineur: based on the International Headache Society classification ICHD-3; experience headache (migraine-like or tension-type-like) on 15+ days/month for 3+ months, and have migraine headaches (either with aura or without aura) on 8+ days/month.
* Participants also must also be classified into a discrepant chronotype: screened using the Morningness/Eveningness Questionnaire, into Definite Morning and Morning types; and Definite Evening and Evening types.

Exclusion Criteria:

* Not classified as a chronic migraineur.
* Not classified into a discrepant chronotype.
* Not classified as low health risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Migraine load difference (evaluated by MIDAS) when exercising in sync with chronotype versus not in sync | Three months
  The Migraine Disability Assessment (MIDAS) is a 5 question assessment which asks participants to recall the number of days activities were affected due to migraine: 1) days of work or school missed, 2) days where productivity at work or school was affected, 3) days not completing housework, 4) days where housework productivity was affected by more than half, 5) days missed family, social, or leisure activities. The assessment will be completed before and after one month of exercise completed in sync with chronotype, and before and after exercise is completed not in sync with chronotype. A one month wash out period will separate these months of exercise.
Migraine load difference (evaluated by HIT-6) when exercising in sync with chronotype versus not in sync | Three months
  The Headache Impact Test (HIT-6) is a 6 question assessment which asks participants to rate on a Likert-type scale (Never, Rarely, Sometimes, Very Often, Always) how activities were affected due to migraine: 1) how often headache pain is severe, 2) how often headache limits usual daily activities, 3) how often you wish you could lie down due to headache, 4) how often you felt too tired due to headaches, 5) how often you felt fed up or irritated due to headache, 6) how often headache limited ability to concentrate on work or daily activities. The assessment will be completed before and after one month of exercise completed in sync with chronotype, and before and after exercise is completed not in sync with chronotype. A one month wash out period will separate these months of exercise.
Migraine load difference (evaluated by MIDAS) when exercising in nature versus indoors | Three months
  The Migraine Disability Assessment (MIDAS) is a 5 question assessment which asks participants to recall the number of days activities were affected due to migraine: 1) days of work or school missed, 2) days where productivity at work or school was affected, 3) days not completing housework, 4) days where housework productivity was affected by more than half, 5) days missed family, social, or leisure activities. The assessment will be completed before and after one month of exercise completed in natural environments, and before and after exercise is completed indoors. A one month wash out period will separate these months of exercise.
Migraine load difference (evaluated by HIT-6) when exercising in nature versus indoors | Three months
  The Headache Impact Test (HIT-6) is a 6 question assessment which asks participants to rate on a Likert-type scale (Never, Rarely, Sometimes, Very Often, Always) how activities were affected due to migraine: 1) how often headache pain is severe, 2) how often headache limits usual daily activities, 3) how often you wish you could lie down due to headache, 4) how often you felt too tired due to headaches, 5) how often you felt fed up or irritated due to headache, 6) how often headache limited ability to concentrate on work or daily activities. The assessment will be completed before and after one month of exercise completed in natural environments, and before and after exercise is completed indoors. A one month wash out period will separate these months of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: James W Navalta, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be available at https://dataverse.harvard.edu/
URL: https://dataverse.harvard.edu/